CLINICAL TRIAL: NCT05746377
Title: Premedication With Metoclopramide in Upper Gastrointestinal Bleeds a Prospective Double Blinded Single Center Randomized Control Trial in a Small Community Hospital
Brief Title: Metoclopramide in Upper Gastrointestinal Bleed
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mercy Health System (Network)
Responsible Party: Principal Investigator, Mudassar Sandozi, Principal Investigator, Mercy Health System
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: #323
Record Dates: First submitted 2023-02-08; First posted 2023-02-27 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Upper GI Bleeding; Bleeds Gastric; Bleed Ulcer; Hemorrhage Gastric; Hemorrhage; Ulcer
Keywords: metoclopramide; prokinetic; Upper endoscopy; EGD; endoscopic gastroduodenoscopy; esophagogastroduodenoscopy
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Hemorrhage; Ulcer | interventions — Metoclopramide; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Randomization protocol instituted by pharmacy, patient and endoscopist blinded to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Metoclopramide (Experimental): Given 10 mg Metoclopramide prior to Endoscopy
  Interventions: Drug: Metoclopramide 10mg
- Placebo (Placebo Comparator): Given saline flush prior to Endoscopy
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Metoclopramide 10mg — IV Metoclopramide
  Other Names: Reglan
  Arms: Metoclopramide
Drug: Saline — Placebo
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to test if metoclopramide can improve effectiveness of endoscopic intervention in upper gastrointestinal (GI) bleeds. The main questions the investigators hope to answer is

Does metoclopramide lessen the need for repeat endoscopy, interventional radiology intervention or surgery in cases of upper GI bleed?

Does metoclopramide improve visibility of the GI walls in cases of upper GI bleed?

DETAILED DESCRIPTION:
The purpose of the study is to see if giving metoclopramide prior to an endoscopy in cases of upper GI bleed can decrease the need for repeat endoscopy due to poor visibility. Metoclopramide stimulates stomach and intestine activity. It is used to treat nausea, vomiting and slow gut movement. The investigators are testing if metoclopramide's effect on stimulating stomach activity can lead to more effective emptying of blood from the stomach and upper intestines in upper GI bleeding so physicians conducting endoscopies can easily see the stomach and intestinal wall and treat the source of bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above
* Admitted to ER or inpatient services at Javon Bea Hospital MercyHealth Riverside
* Present with upper GI bleeding defined as fresh and bright red hematemesis, coffee-ground hematemesis or melena
* Plan to undergo EGD within 24 hours since admission or since first symptoms
* Calculated Glasgow-Blatchford score ≥ 2

Exclusion Criteria:

* Failure to obtain informed consent
* Known allergy to metoclopramide
* Concurrent use of medications known to cause tardive dyskinesia (TD)/extrapyramidal symptoms/neuroleptic malignant syndrome
* History of TD or dystonic reaction to metoclopramide
* Pheochromocytoma, catecholamine-releasing paragangliomas
* Parkinson's Disease
* Epilepsy
* Pregnancy or lactation
* Previous gastrectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-20 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Need for repeat endoscopy, Interventional Radiology Intervention or Surgery due to poor visibility | During Current Hospitalization (up to day 14)
  Will collect if repeat procedure occurred due to poor visibility (True/False)
Toronto Upper Gastroenterology Cleaning Score (TUGS) | During Endoscopy Procedure
  Standardized 0-12 point scale for describing upper gastrointestinal tract visibility, 0 indicating poor visibility, and 12 indicating excellent visibility

SECONDARY OUTCOMES:
Length of Hospital stay (days) | During Current Hospitalization (up to day 14)
  Time in days between admission and discharge
Types of Adverse Neurological Side effects | 3 month f/u
  Dystonia, Akathisia, Parkinsonism, Tardive Dyskinesia, Other
Glasgow-Blatchford Bleeding Score | within 3 hours after admission
  Score from 0-29 estimating risk of gastrointestinal bleed and need for inpatient admission, 0 indicating low risk, 29 indicating high risk of mortality
Endoscopy Findings | During Endoscopy Procedure
  Findings of endoscopy
Endoscopy Start and End Times | During Endoscopy Procedure
  Start and stop times of endoscopies
Number of Blood Units Transfused in 24 hours | within 24 hours after admission
  measure in units of blood transfused

CONTACTS AND LOCATIONS:
Locations (1):
- Javon Bea Hospital-Riverside - MercyHealth, Rockford, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barkun AN, Bardou M, Martel M, Gralnek IM, Sung JJ. Prokinetics in acute upper GI bleeding: a meta-analysis. Gastrointest Endosc. 2010 Dec;72(6):1138-45. doi: 10.1016/j.gie.2010.08.011. PMID 20970794
- [Background] Khan R, Gimpaya N, Vargas JI, Ramkissoon A, Seleq S, Gholami R, Akhtar HJ, Bansal R, Scaffidi MA, Amin S, Bollipo S, Kral J, Lui R, Pawlak KM, Sandhu DS, Bilal M, de-Madaria E, Siau K, Charabaty A, Hashim A, Sanchez-Luna SA, Teshima CW, May GR, Mosko JD, Walsh CM, Grover SC. The Toronto Upper Gastrointestinal Cleaning Score: a prospective validation study. Endoscopy. 2023 Feb;55(2):121-128. doi: 10.1055/a-1865-4180. Epub 2022 May 31. PMID 35642290
- [Background] Daram SR, Garretson R. Erythromycin is preferable to metoclopramide as a prokinetic in acute upper GI bleeding. Gastrointest Endosc. 2011 Jul;74(1):234; author reply 234-5. doi: 10.1016/j.gie.2011.01.059. No abstract available. PMID 21704823
- [Background] Laine L, Barkun AN, Saltzman JR, Martel M, Leontiadis GI. ACG Clinical Guideline: Upper Gastrointestinal and Ulcer Bleeding. Am J Gastroenterol. 2021 May 1;116(5):899-917. doi: 10.14309/ajg.0000000000001245. PMID 33929377
- [Background] Metoclopramide for Acute Upper GI Bleeding - Tabular View - ClinicalTrials.Gov. https://clinicaltrials.gov/ct2/show/record/NCT04771481. Accessed 7 Feb. 2023.